CLINICAL TRIAL: NCT06429917
Title: Impact of Subgingival Instrumentation on Jaw Symptoms of Probable Bruxers Among Patients With Periodontitis- An Interventional Study
Brief Title: Impact of Subgingival Instrumentation on Jaw Symptoms of Probable Bruxers Among Patients With Periodontitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PGIDS/BHRC/24/37
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Periodontitis; Bruxism
Keywords: Inflammation
MeSH Terms: conditions — Periodontitis; Bruxism; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Periodontitis with bruxism (Other): All the participants will undergo subgingival instrumentation with hand scalers, curettes and ultrasonic scaler. Parameters will be recorded at baseline and two, three and six months of time points after subgingival instrumentation.
  Interventions: Other: Subgingival instrumentation

INTERVENTIONS:
Other: Subgingival instrumentation — All the participants will undergo subgingival instrumentation with hand scalers, curettes and ultrasonic scaler. Parameters will be recorded at baseline and two, three and six months of time points after subgingival instrumentation.

SUMMARY:
This study aims to explore the mechanisms by which periodontal disease affects the bruxers and to assess the impact of subgingival instrumentation on jaw symptoms of probable bruxers among patients with periodontitis .

DETAILED DESCRIPTION:
Patients with chronic periodontitis usually describe itching and persistent pain of moderate intensity. Applying masticatory pressure provides relief in these symptoms. However, this practice may lead to the development of bruxism habits in patients over time.

A deeper comprehension of the dynamic interplay between periodontal health and bruxism is crucial for crafting holistic treatment approaches aimed at addressing both symptoms and root causes effectively.

Till now, there has been no report examining the effect of subgingival instrumentation on probable bruxers in periodontitis patients.

. This study aims to assess the impact of subgingival instrumentation on jaw symptoms of probable bruxers in patients with periodontitis

ELIGIBILITY:
Inclusion Criteria:

* 1. Systemically healthy patients 2. Patient having habit of bruxism diagnosed with periodontitis 3. Age between 30-40 years 4. Minimum 20 teeth present in oral cavity

Exclusion Criteria:

1. History of systemic disease such as diabetes or autoimmune disease
2. History of drugs having the potential impact on periodontal status like phenytoin, cyclosporin, calcium-channel blockers or antidepressant drugs.
3. Pregnant or lactating females.
4. Post-menopausal women.
5. Patients diagnosed with temporomandibular disorders- pain and tenderness in the masticatory muscles
6. Patients receiving interventions for bruxism.
7. History of Psychological disorders

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Jaw symptoms | baseline , 2 months , 3 months and 6 months
  Improvement in frequency and intensity of Jaw Symptoms (pain, unpleasantness, sensitivity, tiredness, tension and stiffness) as perceived by the patient.

SECONDARY OUTCOMES:
Bleeding on probing | baseline , 2 months , 3 months and 6 months
  BOP recorded as 1 if bleeding occurs within 15 seconds of probing and 0 (absent) if no bleeding occurred. It will be calculated in %. After adding all the scores, total score will be divided by the total no. of surfaces accessed and multiplied by 100
Gingival index | baseline , 2 months , 3 months and 6 months
  Gingival index by Loe and Silness (1963) will be used to assess severity of gingival inflammation.
Probing pocket depth | baseline , 2 months , 3 months and 6 months
  Probing Pocket Depth (PPD): Probing pocket depth will be measured as the distance from gingival margin to the base of pocket. The probing depth measurements will be assessed using the Periodontal probe. The probe will be inserted in the bottom of pocket and maintained parallel to vertical axis of the tooth. Measurements will be noted at 6sites of a tooth (mesio-buccal, mid-buccal, disto- buccal, mesio-lingual, mid-lingual and disto- lingual). Measurements will be rounded to the nearest whole millimeter.
tooth mobility | baseline , 2 months , 3 months and 6 months
  Tooth mobility is assessed using Miller Mobility Index

CONTACTS AND LOCATIONS:
Overall Officials: VARSHA KAPOOR, BDS, Principal Investigator — PGIDS, ROHTAK
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No